CLINICAL TRIAL: NCT02514525
Title: Multi-center Clinical Study to Evaluate the C2 CryoBalloon Focal Ablation System for the Treatment of Patients With Previously Untreated Dysplastic Barrett's Epithelium
Brief Title: Multi-center Clinical Study to Evaluate the C2 CryoBalloon Focal Ablation System
Acronym: ColdPlayIII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0011
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CryoBalloon Ablation System (Other): Cryoablation treatment of patients with previously untreated (treatment naïve) Barrett's epithelium.
  Interventions: Device: CryoBalloon Ablation System

INTERVENTIONS:
Device: CryoBalloon Ablation System — CryoBalloon Ablation System, a balloon-based cryotherapy device, provides controlled ablation for the treatment of BE. Deployed through the working channel of an endoscope, the Balloon is simultaneously inflated and cooled with an inert cryogen (nitrous oxide) delivered from the handle that ablates the BE cells upon contact with the esophagus.
  Other Names: CryoBalloon Focal Ablation System

SUMMARY:
To evaluate the efficacy and safety of the CryoBalloon Focal Ablation System for the treatment of previously-untreated ("treatment naïve") Barrett's Esophagus (BE)

DETAILED DESCRIPTION:
Coldplay III is a multi-center, prospective study that will provide evidence of the efficacy and safety of the System in treatment of patients with previously untreated (treatment naïve) low grade dysplasia (LGD) or high grade dysplasia (HGD) BE. Subjects may have a maximum of five (5) ablation treatment sessions during their 12 months of study participation to achieve complete eradication of their dysplastic BE and intestinal metaplasia. As many ablations as needed to treat the dysplastic areas are allowed in each treatment session at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Low- or high-grade non-nodular, previously untreated ("treatment naïve") dysplastic BE, confirmed by histopathological analysis. If nodular BE or Intramuscosal Cancer (ImCA) is identified during patient screening, this may be treated with Endoscopic Mucosal Resection (EMR) ≥6 weeks prior to treatment under this protocol. If previous EMR was performed, follow-up endoscopy must be negative for nodular BE. Patients with ImCA must be at low risk for recurrence, confirmed by EMR pathology results negative for positive margin, poorly differentiated carcinoma, and lymphovascular invasion.
* BE length ≤6cm excluding visible BE islands, and Prague Classification C ≥0 / M ≥1
* Older than 18 years of age at time of consent
* Operable per institution's standards
* Provides written informed consent on the approved informed consent form
* Willing and able to comply with study requirements for follow-up

Exclusion Criteria:

* Non-dysplastic or indefinite for dysplasia BE, confirmed by histopathological analysis
* Esophageal stenosis/stricture preventing advancement of a therapeutic endoscope (patients may have the stenosis/stricture dilated and then be treated with CryoBalloon ablation under this protocol at a subsequent procedure ≥2 weeks later)
* Symptomatic untreated strictures
* Any endoscopically-visualized abnormalities such as ulcers, masses or nodules. Neoplastic nodules must first be treated with EMR ≥6 weeks prior to planned treatment under this protocol.
* History of esophageal cancer more extensive than T1a or not meeting criteria for low risk of recurrence (confirmed by EMR pathology results negative for positive margin, poorly differentiated carcinoma, and lymphovascular invasion)
* History of esophageal varices
* Large (>4cm) hiatal hernia
* Prior distal esophagectomy
* Any clinical or histological suspicion of esophageal adenocarcinoma invading into the submucosa by endoscopic mucosal resection (EMR), or confirmed T1a cancer with positive deep margin by EMR
* Active esophagitis grade B or higher
* Severe medical comorbidities precluding endoscopy
* Uncontrolled coagulopathy
* Pregnant or planning to become pregnant during period of study participation
* Patient refuses or is unable to provide written informed consent
* Life expectancy ≤3 years, as judged by the site investigator
* General poor health, multiple co-morbidities placing the patient at risk or otherwise unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2024-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious, CryoBalloon Ablation System-related adverse events | 12 months
Percentage of patients with baseline LGD who have complete eradication of all dysplasia | 12 months
percentage of patients with baseline HGD who have complete eradication of all dysplasia | 12 months
percentage of all treated patients who have complete eradication of all dysplasia (CE-D) | 12 months

SECONDARY OUTCOMES:
Percentage of subjects with complete eradication of all esophageal intestinal metaplasia (CE-IM) | 12 months
Percentage of subjects with progression of dysplasia from LGD to HGD or esophageal cancer, or progression of HGD to cancer | 12 months
  For Baseline LGD and HGD subjects: progression of dysplasia
Incidence of all treatment-related and all serious, non-treatment-related adverse events | 12 months
Incidence of post procedure chest discomfort events / Pain score >0 and <5 | Day 1
  (scored on a 0-10 visual analog pain scale)
Incidence of post procedure chest discomfort events / Pain score ≥5 and requiring narcotic analgesic | Day 7
  (scored on a 0-10 visual analog pain scale)
Mean and Median Pain score on Day 1 post procedure | Day 1
  (scored on a 0-10 visual analog pain scale)
Mean and Median Pain score on Day 7 post procedure | Day 7
  (scored on a 0-10 visual analog pain scale)
Rate of (CE-D) and all esophageal (CE-IM) will be reported as a percentage of all subjects enrolled, and stratified by baseline dysplasia grade | 24 and 36 months
Number of CryoBalloon ablation treatments required to achieve CE-D or CE-IM | 12 months
  (mean and median)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Canto, MD, Principal Investigator — Johns Hopkins Medical Center
Locations (11):
- United States (11):
  - UC Irvine, Orange, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - John Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Manhasset, New York
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Canto MI, Trindade AJ, Abrams J, Rosenblum M, Dumot J, Chak A, Iyer P, Diehl D, Khara HS, Corbett FS, McKinley M, Shin EJ, Waxman I, Infantolino A, Tofani C, Samarasena J, Chang K, Wang B, Goldblum J, Voltaggio L, Montgomery E, Lightdale CJ, Shaheen NJ. Multifocal Cryoballoon Ablation for Eradication of Barrett's Esophagus-Related Neoplasia: A Prospective Multicenter Clinical Trial. Am J Gastroenterol. 2020 Nov;115(11):1879-1890. doi: 10.14309/ajg.0000000000000822. PMID 33156107